CLINICAL TRIAL: NCT01222208
Title: Oral Versus Parenteral Perioperative Nutrition Support to Improve Protein Balance: Stable Isotope Study in Colorectal Surgical Patients
Brief Title: Oral Versus Parenteral Nutrition Support to Improve Protein Balance in Colorectal Surgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Montreal General Hospital (Other); McGill University (Other)
Responsible Party: Principal Investigator, Franco Carli, Dr. Franco Carli, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10-106-GEN
Record Dates: First submitted 2010-10-14; First posted 2010-10-18 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Colon Cancer
Keywords: Bowel resection
MeSH Terms: conditions — Colonic Neoplasms | interventions — Nutritional Status; Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral Nutrition (Active Comparator): Subjects will receive an oral nutrition regimen comprised of 50% of their Resting Energy Expenditure (REE) as dextrose and 20% of their REE as pressurized whey protein
  Interventions: Dietary Supplement: Oral Nutrition with dextrose and pressurized whey protein
- Peripheral Parenteral Nutrition (Placebo Comparator): Subjects will receive a peripheral parenteral nutrition (PPN) regimen comprised of 50% of their Resting Energy Expenditure (REE) as dextrose and 20% of their REE as amino acids.
  Interventions: Dietary Supplement: Peripheral Parenteral Nutrition

INTERVENTIONS:
Dietary Supplement: Oral Nutrition with dextrose and pressurized whey protein — Ten (10) subjects will be randomly assigned to receive an oral nutrition regimen comprised of 50% of their REE as dextrose and 20% of their REE as pressurized whey protein. Subjects will undergo a six-hour stable isotope infusion protocol one day before surgery (to obtain baseline data) and on the first post-operative day. During both infusion protocols, subjects will be asked to carry out their assigned oral nutrition regimen. To minimize fasting during the perioperative period all subjects will receive peripheral parenteral nutrition (PPN) at the time of surgical incision until the first postoperative day.
  Arms: Oral Nutrition
Dietary Supplement: Peripheral Parenteral Nutrition — Ten (10) subjects will be randomly assigned to receive peripheral parenteral nutrition (PPN) regimen comprised of 50% of their REE as dextrose and 20% of their REE as amino acids. Subjects will undergo a six-hour stable isotope infusion protocol one day before surgery (to obtain baseline data) and on the first post-operative day. During both infusion protocols, subjects will be asked to carry out their assigned PPN regimen. To minimize fasting during the perioperative period all subjects will receive PPN at the time of surgical incision until the first postoperative day.
  Arms: Peripheral Parenteral Nutrition

SUMMARY:
A prospective, randomized controlled study, using stable isotope methodology, is proposed to determine whether an oral nutrition support regimen, containing pressurized whey protein and glucose, is more effective at normalizing the metabolic response to surgery than a standard peripheral parenteral nutrition (PPN) support regimen, containing amino acids and glucose, in colorectal surgical patients studied before and after surgery. The effectiveness of the nutrition support regimens will be determined by: whole body protein balance, synthesis rates of hepatic secretory proteins, resting energy expenditure and substrate utilization, as well as circulating metabolites concentrations.

ELIGIBILITY:
Inclusion Criteria:

1. The American Society of Anesthesiologists' (ASA) class 1 to 3
2. Colorectal surgery for non-metastatic disease (including right, transverse, left, sigmoid, subtotal, total, and hemicolectomy)
3. Nutrition status: 18.5 < body mass index < 30 kg/m2, stable weight over the preceding three months (< 10% body weight loss), serum albumin > 35g/l

Exclusion Criteria:

1. History of hepatic failure (Child-Pugh score A-C and transaminases outside the normal range)
2. Renal impairment (Serum Creatinine outside normal range)
3. Cardiac failure (New York Heart Association (NYHA) classes I-IV)
4. Hepatic, Renal, Cardiac transplant
5. Endocrine disorders: diabetes type I & II, hyper and hypothyroidism
6. Active inflammatory bowel or diverticular disease (Crohn's Disease, Ulcerative Colitis)
7. Musculoskeletal or neuromuscular disease
8. Anemia defined as hematocrit < 30, hemoglobin < 10 g/dl, albumin < 25 mg/dl
9. Previous spine surgery or scoliosis limiting use of epidural
10. Pregnancy
11. Use of Steroids
12. Milk protein allergy or intolerance

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-03; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Whole body protein balance | 1 year
  Whole body protein balance (the difference between protein synthesis and protein breakdown) as assessed by the kinetics of a stable, non-radioactive, isotope tracer infusion of L-[1-13C] leucine

SECONDARY OUTCOMES:
Synthesis rates of hepatic secretory proteins | 1 year
  Synthesis rates of hepatic secretory proteins, including the classically positive acute phase reactant fibrinogen and the classically negative acute phase reactant albumin, as assessed by incorporation of the stable, non-radioactive, isotope tracer L-[2H5] phenylalanine into plasma Very Low Density Lipoprotein ApolipoproteinB100.

CONTACTS AND LOCATIONS:
Overall Officials: Franco Carli, M.D., Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Result] Schricker T, Meterissian S, Lattermann R, Adegoke OA, Marliss EB, Mazza L, Eberhart L, Carli F, Nitschman E, Wykes L. Anticatabolic effects of avoiding preoperative fasting by intravenous hypocaloric nutrition: a randomized clinical trial. Ann Surg. 2008 Dec;248(6):1051-9. doi: 10.1097/SLA.0b013e31818842d8. PMID 19092350